CLINICAL TRIAL: NCT05359562
Title: Harnessing Hormonal Variation to Probe Neural Mechanisms and Optimize CBT Outcomes for OCD
Brief Title: How Hormones and Exposure and Response Prevention (EX/RP) Affect the Brain of People With OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: New York State Psychiatric Institute (Other); New York University (Other); Research Foundation for Mental Hygiene, Inc. / Columbia University (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01MH121608-01A1 (NIH); 1R01MH121597-01A1 (NIH)
Record Dates: First submitted 2022-04-28; First posted 2022-05-04 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: OCD
Keywords: OCD; Exposure and Ritual Prevention; Extinction Learning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study hypotheses will be masked to participant, therapist, and outcome assessor. Assignment of women participants to groups will be masked to therapist, investigator, and outcome assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator (Active Comparator): Male participants will receive a brief EX/RP protocol within a 10-day window.
  Interventions: Behavioral: Exposure & Response Prevention (EX/RP)
- Experimental 1 (Experimental): Half of female participants will be randomized to receive a brief EX/RP protocol within the first 10 days after the start of menstruation (early follicular phase).
  Interventions: Behavioral: Exposure & Response Prevention (EX/RP)
- Experimental 2 (Experimental): Half of female participants will be randomized to receive a brief EX/RP protocol in days 12-22 of the menstrual cycle (late follicular, early luteal phase).
  Interventions: Behavioral: Exposure & Response Prevention (EX/RP)

INTERVENTIONS:
Behavioral: Exposure & Response Prevention (EX/RP) — Exposure and Response Prevention (EX/RP) is a type of Cognitive Behavioral Treatment for treating OCD. This is a brief protocol consisting of 8 sessions of exposure and Response Prevention (EX/RP). This protocol includes two psychoeducation/planning sessions, followed by six exposure sessions.

SUMMARY:
Studies show that hormones affect the brain's fear extinction network, which is relevant for therapy involving exposure and response prevention (EX/RP), a first-line treatment for obsessive compulsive disorder (OCD). This study will examine the effect of delivering EX/RP to women during different phases in their menstrual cycle to determine the effects of hormones on the fear extinction network and on their OCD symptoms.

DETAILED DESCRIPTION:
This study involves neuroimaging and a brief EX/RP protocol. The investigators will recruit both male and female participants. All participants will complete neuroimaging, hormonal assays and symptom ratings before and after a brief course of EX/RP. Female participants will be randomized to complete brief EX/RP during distinct phases of their menstrual cycles. This design will allow the investigators to study the effects of hormonal variation during the menstrual cycle and sex on the fear extinction network and on EX/RP outcome. The long-term goal is to optimize EX/RP for individuals suffering from OCD. Men will also be recruited for this study to further explore biological sex differences. The results will elucidate treatment mechanisms and could lead to personalized treatment recommendations for women with OCD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic and Statistical Manual of Mental Disorders (DSM-5) Diagnosis of OCD;
2. Male and female subjects aged between 18- 45;
3. Women must be menstruating and regularly cycling
4. Ability to tolerate a treatment-free period;
5. No psychotropic medication in the past 12 weeks
6. At entry, at least moderate severity OCD
7. Willingness and ability to give written informed consent after full explanation of study procedures.

Exclusion Criteria:

1. Use of birth control (oral contraception or IUD) that affects the menstrual cycle, or menopause.
2. Pregnancy. Women of childbearing potential will be required to sign a statement indicating their intention to avoid pregnancy during the study.
3. Neurologic or medical condition that would prevent safe participation in the full study protocol.
4. Any contradiction to magnetic resonance imaging (e.g., metallic implants or devices).
5. Comorbid psychiatric conditions that significantly elevate the risks associated with study participation or confound results.
6. Patients with prominent suicidal ideation or with a recent suicide attempt.
7. Current psychotherapy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
fMRI | Baseline to approximately 4 weeks later
  Slope of change in brain activation (fMRI)
OCD Symptoms | Baseline to approximately 4 weeks later
  Slope of change in Obsessive Compulsive Symptom Severity (Yale-Brown Obsessive Compulsive Scale)

SECONDARY OUTCOMES:
rs fMRI | Baseline to approximately 4 weeks later
  Slope of change in resting state functional connectivity (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Edna B Foa, PhD, Principal Investigator — University of Pennsylvania; Helen B Simpson, MD, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania